CLINICAL TRIAL: NCT01875926
Title: Phase I, Single-centre, Open-label Study to Evaluate the Pharmacokinetics of ALX-0171, Administered by Oral Inhalation or Intravenously, in Healthy Male Volunteers
Brief Title: ALX-0171 Phase I Pharmacokinetic Study in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALX-0171-1.3/13; 2013-001425-71 (EudraCT Number)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Healthy; RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — gontivimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ALX-0171 Oral Inhalation - Single Dose (SD) (Experimental)
  Interventions: Biological: ALX-0171
- ALX-0171 Oral Inhalation - Multiple Dose (MD) (Experimental)
  Interventions: Biological: ALX-0171
- ALX-0171 Intravenous (IV) (Experimental)
  Interventions: Biological: ALX-0171

INTERVENTIONS:
Biological: ALX-0171 — single dose of 200 mg ALX-0171 via oral inhalation
  Arms: ALX-0171 Oral Inhalation - Single Dose (SD)
Biological: ALX-0171 — repeated doses of 200 mg ALX-0171 via oral inhalation once daily for 5 consecutive days
  Arms: ALX-0171 Oral Inhalation - Multiple Dose (MD)
Biological: ALX-0171 — Single dose of 0.3 mg/kg body weight ALX-0171 via intravenous administration
  Arms: ALX-0171 Intravenous (IV)

SUMMARY:
The overall aims of the study are:

* To provide additional information on the pharmacokinetics of ALX-0171 by measuring (i) local (bronchoalveolar lavage fluid (BALF)) and systemic (plasma) concentrations of ALX-0171 after oral inhalation, and (ii) systemic (plasma) and urine concentrations after intravenous administration.
* To further determine the safety and local and systemic tolerability of ALX-0171.
* To further evaluate local (induced sputum) and/or systemic (serum) immunogenicity of ALX-0171, by analysing the potential occurrence of anti-drug antibodies (ADA).

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking healthy male volunteers, (18-55 years, extremes included).
2. Good health condition, as determined by medical history, physical examination and clinical laboratory testing
3. Body mass index (BMI) within normal range: 18.0 ≤ BMI < 30.0 (kg/m2)
4. Haematology and chemistry parameters within normal range, or showing no clinically relevant deviations (as judged by the Investigator)
5. Heart rate and/or blood pressure within normal range (as judged by the Investigator)
6. Electrocardiogram (ECG) within normal range, or showing no clinically relevant deviations (as judged by the Investigator)
7. Negative urine test for selected drugs of abuse at screening
8. Negative alcohol breath test upon check-in at study unit
9. Negative hepatitis panel (including hepatitis B surface antigen (HBsAg) and anti-hepatitis C virus antibodies (anti-HCV)), and negative human immunodeficiency virus (HIV) antibody screens
10. Willingness to consent to using an effective contraceptive method (by using 2 methods of contraception in combination with a female partner: at least 1 of the contraception methods must be a barrier contraception method, e.g., condom) during the study and for at least 3 months after last study drug administration
11. Ability to comprehend and willingness to sign an Informed Consent Form (ICF)

    For oral inhalation only:
12. Lung function test which shows a Forced Expiratory Volume in 1 second (FEV1) ≥ 90% of predicted value
13. Ability to retro-breathe with nebulizer
14. Height between 170 and 190 cm (extremes included)
15. Ability to produce a sufficient amount of induced sputum (at least 400 μL containing visual sputum plugs) to assess immunogenicity

Exclusion Criteria:

1. Current smokers, or ex-smokers abstinent from tobacco for less than one year, or a history of smoking more than 10 packs a year
2. Symptomatic viral infection, or suspicion thereof (including rhinitis) in the last 14 days prior to dosing
3. Signs of active pulmonary infection or other pulmonary inflammatory conditions, even in the absence of febrile episodes, in the last 14 days prior to dosing
4. History or presence of disease in the kidneys and/or heart, lungs, liver, gastrointestinal tract, endocrine organs or other conditions such as metabolic disease known to interfere with the absorption, distribution, metabolism or excretion of drugs
5. Malignancy, or prior malignancy, with a disease-free interval of < 5 years after diagnosis and intervention, except basal cell carcinoma (treated curatively)
6. Autoimmune disorders such as (but not limited to) lupus erythematosus, multiple sclerosis, rheumatoid arthritis, or sarcoidosis.
7. History of hypersensitivity or allergies to any drug compound, including constituents of ALX-0171
8. History of previous administration of ALX-0171, or any other inhaled biologic or drug targeting the Respiratory Syncytial Virus (RSV) F protein. In any other case of use of biologics: at least 6 months before administration of first study medication, or the time of duration of the pharmacodynamic effect, or 10 times the half-life of the respective drug, whatever is longer
9. Receipt of any investigational drug within 60 days prior to dosing
10. Intake of prescribed or over-the-counter medication within 14 days prior to dosing (≤ 3 g/day paracetamol is allowed)
11. History or presence of alcohol or drug abuse
12. Blood donation (> 500 mL) or a comparable blood loss within three months prior to dosing
13. Planned donation of germ cells, blood, organs, bone marrow during the course of the study or within 6 months thereafter
14. Any other condition or prior therapy which, in the opinion of the Investigator, would make the subject unsuitable for this study
15. Vulnerable subjects (e.g., persons kept in detention)

    For oral inhalation only:
16. History or presence of atopy or any condition associated with airway hyperresponsiveness (e.g., allergic or non-allergic asthma, chronic obstructive pulmonary disease (COPD))
17. FEV1 drop of > 10% after inhalation of 4 mL of ALX-0171 placebo (measured at 5 min after the end of inhalation)
18. Contra-indication for sputum induction, such as (but not limited to) recent eye surgery, recent fractured ribs and recent (or history of) pneumothorax

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: concentration of ALX-0171 after oral inhalation in BALF samples and in plasma samples | Day 1 to Day 9
Pharmacokinetics: ALX-0171 concentration in plasma and urine after intravenous administration | Day 1 to Day 4

SECONDARY OUTCOMES:
Safety and tolerability: safety markers | from signing of Informed Consent Form (ICF) until last follow-up visit (i.e 35 to 42 days after first study drug administration)
  * Lung function test pre- and post-inhalation with 4 mL of ALX-0171 placebo (on Day -1, applicable for oral inhalation only).
  * Lung function tests
  * Physical examination (including physical examination of the lung for oral inhalation)
  * Vital signs
  * 12-lead ECG.
  * Clinical laboratory
  * Limited safety lab (haematology + limited chemistry).
  * Adverse events (AEs) and concomitant medication
Immunogenicity: concentration of Anti-Drug Antibodies (ADA)in induced sputum (after oral inhalation only) and serum | during screening until last follow-up visit (i.e. 35 to 42 days after first study drug administration)

CONTACTS AND LOCATIONS:
Overall Officials: Steven De Bruyn, MD, Study Director — Ablynx NV
Locations (1):
- Antwerp, Belgium